CLINICAL TRIAL: NCT03924167
Title: The Weaving Healthy Families Program to Promote Wellness and Resilience and Prevent Alcohol and Other Drug Abuse and Violence
Brief Title: The Weaving Healthy Families Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Catherine E. McKinley, Associate Professor, Tulane University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-1372; 5R01AA028201-03 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Abuse; Drug Use; Violence, Domestic; Child Abuse; Diet Modification; Health Behavior; Health Knowledge, Attitudes, Practice; Relationship, Family; Relation, Parent-Child; Emotional Stress
MeSH Terms: conditions — Alcoholism; Health Behavior; Behavior; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The proposed research will use a stepped-wedge trial design (SWTD) to test the efficacy of a culturally modified intervention that is facilitated by Tribally-based community health representatives (CHRs) and the consolidated framework for implementation research (CFIR) to examine the barriers and facilitators for intervention sustainability and implementation.
Who Masked: Participant, Care Provider
Masking Description: Families and CHRs will be blinded to the order they receive the intervention and notified a month in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Families Receiving Weaving Healthy Families Intervention (Experimental): The Weaving Healthy Families curriculum is a cognitive-behavioral, support group model for high-risk families related to alcohol, tobacco, or other drugs (ATOD) and/or or domestic violence, child abuse, or neglect. This curriculum is tailored for all ages (i.e., (a) parents/caregivers; (b) early childhood (5-7); (c) children (8-11); and (d) adolescent (12-17) and is aimed at reducing alcohol and other drug (AOD) abuse, promote unity, address mental health problems, strengthen parenting skills, and bolster wellness and resilience.
  Interventions: Behavioral: Weaving Healthy Families Program
- Families who have not yet receive the Weaving Healthy Families (No Intervention): Baseline group --data will be collected prior to receiving the intervention in this stepped-wedge trial design.

INTERVENTIONS:
Behavioral: Weaving Healthy Families Program — The Weaving Healthy Families program is created from integrating the widely disseminated, ecological, innovative, and culturally grounded Framework of Historical Oppression, Resilience, and Transcendence (FHORT) with the the Celebrating Families! evidenced-based program (EBP). The goal of this program is to reduce and postpone Alcohol and other Drug (AOD) use, decrease and prevent violence in families, and promote resilience and wellness (including mental health) among NA adults and youth. This intervention seeks to promote wellness by targeting key behavioral (AOD), mental/emotional (emotional regulation/anger management, cognitions, resilience), social and familial (healthy and safe relationships, the family environment, and parenting), cultural (values, traditions), and physical (nutrition) factors.
  Other Names: Celebrating Families! Program
  Arms: Families Receiving Weaving Healthy Families Intervention

SUMMARY:
Alcohol and other drug (AOD) abuse and violence in families are co-occurring risk factors that drive health disparities and mortality among Native Americans (NA), making the long-term goal of this research is to promote health and wellness, while preventing and reducing AOD abuse and violence in NA families by testing an efficacious, sustainable, culturally-relevant and family-centered intervention for cross-national dissemination. The central hypothesis is that the sustainable and community-based Weaving Healthy Families program, will reduce and postpone AOD use among NA adults and youth, decrease and prevent violence in families, and promote resilience and wellness (including mental health) among NA adults and youth. The expected outcomes of the proposed research are an efficacious, culturally relevant, and sustainable community based program to promote health and wellness that will address the factors that drive health disparities and promote individual, family, and community resilience.

DETAILED DESCRIPTION:
Alcohol and drug (AOD) abuse and family violence are co-occurring risk factors for Native American (NA) health disparities and are associated with the leading causes of death, such as cardiovascular disease (CVD) and diabetes. However, extant interventions often fail to holistically promote resilience, health, and wellness and instead address problems in isolation. There have been few NA culturally-based and family-focused, interventions that enhance family resilience and prevent and reduce AOD abuse and violence in families. Given the gap in community and culturally-grounded programs to prevent AOD abuse and violence in families, there is a critical need to test the efficacy of such sustainable community-based interventions. The long-term goal of this research is to promote health and wellness, while preventing and reducing AOD abuse and violence in NA families by testing an efficacious, sustainable, culturally-relevant and family-centered intervention for cross-national dissemination. Using community-based participatory research methods (CBPR), the overall objectives of the proposed research is to use a stepped-wedge trial design (SWTD) to test the efficacy of a culturally modified intervention that is facilitated by Tribally-based community health representatives (CHRs) and to use the consolidated framework for implementation research (CFIR) to examine the barriers and facilitators for intervention sustainability and implementation. The central hypothesis is that the sustainable and community-based, "Weaving Healthy Families program"-a shortened and culturally adapted version of the Celebrating Families! Program-will reduce and postpone AOD use, decrease and prevent violence in families, and promote resilience and wellness (including mental health) among NA adults and youth. This intervention seeks to promote wellness by targeting key behavioral (AOD), mental/emotional (emotional regulation/anger management, cognitions, resilience), social and familial (healthy and safe relationships, the family environment, and parenting), cultural (values, traditions), and physical (nutrition) factors. Investigators test the efficacy and gain knowledge in sustainability and implementation by: Aim 1: Test the efficacy of the modified intervention on AOD and violence reduction and resilience enhancement. Using an open cohort, multiple baseline SWTD and multilevel and longitudinal modeling, investigators will test our working hypothesis that the intervention will reduce parental AOD misuse and violence, postpone youth AOD use, and enhance family members' resilience and wellness. Aim 2: Evaluate the sustainability and feasibility of the intervention's implementation. Investigators will use the CFIR and a convergent mixed-method design to evaluate barriers and facilitators to intervention implementation, testing our working hypothesis that the modified intervention will provide a culturally relevant and feasible model to promote wellness in a sustainable way. The expected outcomes of the proposed research are an efficacious, culturally relevant, and sustainable community based program to promote health and wellness for tribes cross-nationally.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for community health representatives (CHR)s.

   1. 18 years of age or older
   2. have at least a high school degree
   3. have experience and/or interest in working with tribal children and families.
2. Exclusion criteria:

   1. having less than a high school degree
   2. not having experience with tribal families
3. Inclusion criteria for families

   1. includes written consent for adults and assent for children ages 12-17.
   2. at least one parent/caregiver who is a member of the focal tribe and at least one child, aged 12-18 living in the household
4. Exclusion Criteria:

   1. current protective order
   2. current intimate partner violence (IPV) record will be excluded.

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in the AUDIT= Alcohol Use Disorders Identification Test | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  The 10-item AUDIT identifies alcohol consumption, drinking behaviors, and alcohol-related problems among adults. Scores for each question range from 0 to 4, with the first response for each question (eg never) scoring 0, the second (eg less than monthly) scoring 1, the third (eg monthly) scoring 2, the fourth (eg weekly) scoring 3, and the last response (eg. daily or almost daily) scoring 4. For questions 9 and 10, which only have three response, the scoring is 0, 2 and 4 (from left to right). A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Change in the DAST= Drug Abuse Screening Test | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  A 10-item form used to assess drug use with adults. Participants receive 1 point for every "yes" answer with the exception of question #3, for which a "no" answer receives 1 point.
  Degree of problems by score: 0=no problems reported, 1-2 = low level, 3-5=moderate level, 6-8=substantial level, 9-10=severe level.
Change in the AADIS= Adolescent Alcohol and Drug Involvement Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Adolescent alcohol and other drug (AOD) use will be assessed using the AADIS, which assesses frequency of AOD as well as 14 items assessing severity of AOD misuse. Scores are added with results indicating: Scores of 0 = No alcohol or other drug use. Scores of 1-36 = Alcohol and/or other drug use present, does not reach threshold for substance use disorder based on DSM-IV criteria. Scores of 37 or higher = Alcohol and/or other drug use present which may reach DSM IV criteria.
Change in the CRAFFT=Car, Relax, Alone, Forget, Friends, Trouble | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  A 9-item evidenced-based screening tool, will be used to assess AOD misuse, (alcohol and drug use separately and holistically). 9 items. 1-3 number of days used substances. 4-9 yes, no responses with each "yes" response scoring 1 point. A total score of 2 or higher is a positive screen, indicating a need for additional assessment.
Change in the FES=Family Environment Scale-Short Form | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Assesses key components of healthy functioning through the following subscales: cohesion, expressiveness, conflict, independence, achievement orientation, intellectual and cultural orientation, active-recreational orientation, moral-religious emphasis, organization, and control. 90 item scale. Respondents mark whether each item is true (1) = 1 or false (2) =0 for them. Scoring: To determine a person's raw score (RS), count the number of responses in each subscale, and enter the total in the RS box at the bottom. Scores range from 0-10 for each subscale, with higher scores indicating higher levels of that construct. To determine the family's mean RS for each subscale, average the subscale raw scores for all members of that family.
Change in the FRI=Family Resilience Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Assesses family resilience in current family and family of origin. Scoring: Add responses for each item. Total scores range from 0-20, with higher scores indicating a higher degree family resilience. Each of the items can be thought of as a protective factor, cumulatively contributing to the holistic measure of family resilience.
Change in the CD-RISC=Conner-Davidson Resilience Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Assesses individual or psychological resilience. 10-item scale. Scoring of the scale is based on summing the total of all items, each of which is scored from 0-4. For the CD-RISC-10, the total score ranges from 0-40. Higher scores indicate higher levels of psychological resilience.
Change in the CTS-2=Conflict Tactics Scale 2 | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  The CTS2 is a comprehensive self-reported inventory designed to measure five scales: Negotiation (positive verbal conflict resolution skills), Psychological Aggression, Physical Assault, Sexual Coercion, and Injury. Respondents rate each item on a 7-point Likert- style frequency scale (0 = this has never happened before, 1 = once in the past year, 2 = twice in the past year, 3 = 3-5 time in the past year, 4 = 6-10 times in the past year, 5 = 11-20 times in the past year, 6 = more than 20 times in the past year, and 7 = not in the past year, but it did happen before). To create interpretable scores, values 1 and 2 remained the same, and values 3 through 6 were recoded to be the midpoints (3 = 4, 4 = 8, 5 = 15, 6 = 25). Frequency scores (how often) for each subscale are added (Range 1-12 for frequency, higher scores indicating higher levels of each subscale). Dummy are created with each item and subscale for prevalence (1=yes in the past year; 0=not in the past year).
Change in the DAS-SF/DAS-C= Dysfunctional Attitudes Scale-Short Form/Child | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Assesses dysfunctional attitudes, which have been shown to be precursors to depression and stress. Items are on a 4-point Likert scale (1-Totally agree to 4-Totally disagree). Items should be scored so that total score reflects greater dysfunctional attitudes. This means that most items will be reverse coded. Subtracting 5 from an item score will reverse score that item. Items are on a 4-point Likert scale (1-Totally agree to 4-Totally disagree).
Change in the SWLS=Satisfaction with Life Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  A short measure of life satisfaction. The SWLS is a five-item scale designed to measure global judgements about one's life satisfaction. Respondents indicated how much they agreed or disagreed with each of the five items using a seven-point scale that ranged from 'strongly disagree' to 'strongly agree'. The summed scale ranged from 5-35, with higher scores indicating greater life satisfaction.
Change in the DERS-18= Difficulties in Emotional Regulation Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  An 18-item measure of emotional regulation and anger management. Sum items for each subscale with Items 1, 4, and 6 being reverse-coded. Add subscale totals for the total summative scale as follows: Awareness (# 1, 4, 6); Clarity (#2, 3, 5); Goals (#8, 12, 15); Impulse (#9, 16, 18); Nonacceptance (#7, 13, 14), and Strategies (#10, 11, 17).
Change in the BRFSS=Behavioral Risk Factor Surveillance System | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Items taken from the BRFSS on the modules on chronic health, diet, and exercise. Subscales/items: CDC HRQOL- 4-Physical health, mental health, days not good, 4 items. Scoring: To obtain this estimate, responses to questions 2 and 3 are combined to calculate a summary index of overall unhealthy days, with a logical maximum of 30 unhealthy days. Participants were asked whether they had any of 16 chronic health problems (1 yes, 2 no). Scored to create overall measure of health problems. Four diet questions about frequency of consuming. Summed to create mean scores for each item. 4 individual exercise-related questions, individually scored. 4-item HDCM BRFSS (Past 30 days, health-related problems). Score summed. With the exception of the full of energy item, higher scores indicate poorer health.
Alabama Parenting Questionnaire-9/ APQ-SF | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), 6, 9, and 12 month follow-ups.
  Measures five dimensions of parenting. 13-item scale. Items (e.g. You threaten to punish your child and then do not actually punish him/her) are rated on a 5 point Likert Scale (1 = never; 2 = almost never; 3 = sometimes; 4 = often; 5 = always). Higher scores indicate higher ratings of the measured parenting practice (i.e. Positive Parenting, Inconsistent Discipline, Poor Supervision).

SECONDARY OUTCOMES:
Change in the CSAP = Center for Substance Abuse Prevention (Minority Initiative) | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Secondary measures of AOD abuse among youth and adults. 41 items answered on likert-type scales, which are summed and averaged.
Change in the PSDQ-SF=Parenting Styles and Dimensions Questionnaire-Short Form | Change from Baseline, Pre-test, and Post-test (within one month of completion of intervention).
  Measure of parenting styles, which are associated with more optimum and less optimum parent-child relationships. 124-item scale. There are 27 items in the Authoritative Construct with the following subscales: Warmth and Involvement, Reasoning and Induction, Democratic Participation, and Good Natured/Easy Going. There are 20 items for the Authoritarian Construct with the following subscales: Verbal Hostility, Corporal Punishment , Non-reasoning, Punitive Strategies, and Directiveness. There are 15 items for the Permissive Construct with the following subscales: Lack of Follow Through, Ignoring Misbehavior, and Self Confidence. Each item of the scale were evaluated with the five points likert described as, "never" (1) to "always" (5) . Scores for each authoritarian, authoritative, and permissive parenting styles are achieved by creating the mean for each construct with higher scores indicating higher levels of the given construct (Ranging from 1-5).
Change in the SRHP=Self-Rated Health Practices | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of health self-efficacy. The 28-item Self-Rated Abilities for Health Practices Scale (SRHP), which is a 5-point scale ("not at all" = 0 to "completely" = 4) to measure perceived ability to implement health promoting behavior. Scores range from 0-112, with higher scores indicating greater health practices self-efficacy.
Change in the Kidscreen | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of health self-efficacy among youth. 27 items. Items are summed and/or means are calculated for a total health-related quality of life.
Change in the GAD-7=Generalized Anxiety Disorder | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of anxiety symptoms for adults. This seven-item, self-report questionnaire focused on symptoms of feeling nervous, anxious or on edge, not being able to stop or control worrying, and having trouble relaxing. Respondents rated the how often they experienced these symptoms over the past two weeks (0 = not at all, 3 = nearly every day). Scores ranged from 0-21 with higher scores indicating more severe symptoms.
Change in the SCARED=Screen for Child Anxiety Related Emotional Disorders | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of anxiety symptoms for youth. 41-item scale. Responses range from 1=Not True or Hardly Ever True to 3=Very True or Very Often True. Items are summed to form a total score. Scores range from 41-123. Higher scores indicated higher levels of anxiety related symptomatology. A score of 25 or greater is indicative of the presence of an anxiety disorder. Scale include subscales with scores in parenthesis for each indicative of levels of clinical significance for School Avoidance (3), Social Anxiety Disorder (8), Separation Anxiety Disorder (5), Panic Disorder (7), and Significant Somatic Symptoms (7).
Change in the PHQ-9= Patient Health Questionnaire | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of depressive symptoms for adults. Participant's indicate how often over the past two weeks they were bothered by depressive symptoms. For each of the nine items, four response options were available. These were: 0 = 'not at all', 1 = 'several days', 2 = 'more than half the days', and 3 = 'nearly every day'. When summed, the nine scale items had a possible range of 0 to 27 and the total score corresponded to an individual's level of depressive symptoms along a continuum that was scored as: minimal (score of 0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27) depression. PHQ-9 scores of 10 or higher indicate clinical depression, a cut point validated across numerous studies.
Change in the PC-PTSD=Primary Care PTSD Screen | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of PTSD for adults. Preliminary results from validation studies suggest that a cut-point of 3 on the PC-PTSD-5 (e.g., respondent answers "yes" to any 3 of 5 questions about how the traumatic event(s) have affected them over the past month) is optimally sensitive to probable PTSD. Optimizing sensitivity minimizes false negative screen results. Using a cut-point of 4 is considered optimally efficient. Optimizing efficiency balances false positive and false negative results.
Change in the C-SSRS=Columbia-Suicide Severity Rating Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of suicide symptoms for adults. Add symptoms of suicidal ideation (0/1). Any score greater than 0 indicates some level of suicide ideation. A score of 4 (active suicidal ideation with some intent to act) or 5 (active suicidal ideation with specific plan and intent) on suicidal ideation indicate serious suicidal ideation.
Change in the SHALOM= Spiritual Health and Life-Orientation Measure | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of spiritual health and wellness. Spiritual well-being is assessed using the Spiritual Health and Life-Orientation Measure (SHALOM), which is a 42-item scale. Calculate mean scores for each of the 4 domains. Difference between the ideals and lived experience scores can be used to investigate the level of spiritual harmony or dissonance. Includes two additional questions (importance of religion, importance of spirituality) which should be scored separately. Item responses range from 1 (very low) to 5 (very high). These are added and an overall mean is created, with higher scores indicating higher spiritual well-being.
Change in Communal Mastery Scale | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of community resilience and cohesion. 10-item scale. Items were summed to find total scores of communal mastery. Total scores range from 10 to 40 with higher scores indicating more community resilience and cohesion (a more optimum outcome).
Change in the SSI=Social Support Index | Change from Baseline, Pre-test, Post-test (within one month of completion of intervention), and 12 month follow-ups.
  Measure of social, familial, and community support. The 17 items are coded as follows: 1 Strongly disagree; 2 Disagree; 3 Neutral; 4 Agree; or 5 Strongly Agree. Scores are added to indicate levels of social and familial support (higher scores, higher support). Some items (7, 9, 10, 14, 17) are reversed coded.
Change in the IGI=In-Group Identification | Change from Baseline, Pre-test, and Post-test (within one month of completion of intervention).
  Measure of ethnic identity. Measure mean score across items.
Change in the HOS=Historical Oppression Scale | Change from Baseline, Pre-test, and Post-test (within one month of completion of intervention).
  Measure of perceived historical oppression. Add responses for each item. Total scores range from 10-50, with higher scores indicating a higher degree of reported historical oppression.
Change in the HLS=Historical Loss Scale-R | Change from Baseline, Pre-test, and Post-test (within one month of completion of intervention).
  Measure of perceived historical loss. The Historical Loss Scale (HLS) is an adapted version, creating a 15 time scale measuring the frequency with which people think of historical loss from a continuum of the following: 1 = 'several times a day'; 2 = 'daily'; 3 = 'weekly'; 4 = 'monthly'; 5 = 'yearly or at special times'; and 6 = 'never'. The following items were added the following culturally relevant items to the original 12-item scale: "Loss of family unity and increase in family violence"; "Loss of respect for women"; and "Losses from man-made disasters, flooding, pollution, and destruction of natural resources." Responses were summed (range = 15-75) and higher values indicated a higher degree of historical loss.
Change in the EDS=Everyday Discrimination Scale | Change from Baseline, Pre-test, and Post-test (within one month of completion of intervention).
  Measure of perceived discrimination. This 5-item scale measures the frequency 5 (every day) to 0 (never) that people experience discrimination, with higher scores indicating greater perceived discrimination.
Change in the ACE=Adverse Childhood Experiences | Change from Baseline, Pre-test, and Post-test (within one month of completion of intervention).
  Measure of child maltreatment and childhood stress and trauma. Yes/no items are added indicating total numbers of adverse childhood events. Higher scores more adverse experiences.
Change in the ICBS= Implementation Citizenship Behavior Scale | Change from from Baseline and 12 Month Follow-up.
  Measure of facilitator behaviors and attitudes about the intervention. The six items of this scale are added (0=not at all to 5=frequently if not always) with higher scores indicating higher levels of practitioners exceeding expected job tasks.
Change in the Intervention AS-36= Evidence-based Practice Attitude Scale | Change from from Baseline and 12 Month Follow-up.
  Measure of consolidated framework for implementation research. Items for this 36-item scale are added with 0=not at all to 5-very great extent, with higher scores indicating the better fit for this intervention.
Change in the PSI=Program Sustainability Index | Change from from Baseline and 12 Month Follow-up.
  Measure of Program Sustainability. Items are added from 0=not at all true to 2=very much true for an overall measure of program sustainability.

CONTACTS AND LOCATIONS:
Locations (1):
- Catherine McKinley, New Orleans, Louisiana, United States